CLINICAL TRIAL: NCT06245421
Title: Multicentric, Randomized, Comparative Clinical Study on the Evaluation of the Efficacy and Safety of DM934 Versus Théalose on the Treatment of Moderate to Severe Ocular Dryness
Brief Title: Evaluation of the Efficacy and Safety of DM934 Versus Théalose on Eye Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus Pharma (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23E0548
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (Experimental)
  Interventions: Device: DM934
- Comparator (Active Comparator)
  Interventions: Device: Théalose

INTERVENTIONS:
Device: DM934 — 1 drop in each eye, 4 to 6 times per day
  Arms: Investigational product
Device: Théalose — 1 drop in each eye, 4 to 6 times per day
  Arms: Comparator

SUMMARY:
This study is a multicentric, comparative, randomized, investigator-blinded, parallel group study to demonstrate the non-inferiority of DM934 in comparison with Théalose in terms of cornea and conjunctiva staining (Oxford score) on patients with moderate to severe ocular dryness, after 35 days of treatment

ELIGIBILITY:
Inclusion Criteria:

* Subject with a moderate to severe dry eye syndrome needing artificial tears in the 3 months preceding the inclusion.
* Subject having used only artificial tears without preservative (NaCl 0.9%, Larmabak®) during 1 to 2 weeks before inclusion (up to 6 times a day) (given during wash-out period).
* Subject with a score ≥ 18 for the OSDI (Ocular Surface Disease Index).
* Subject with at least one eye with:

  * Global ocular staining (cornea and conjunctiva) ≥4 and ≤9 on the Oxford scale (0 to 15)

AND one of the following criteria:

* Schirmer test ≥ 3 mm/5 min and ≤ 9 mm/5 min OR
* Sum of 3 measurements of Tear film Break-Up Time (TBUT) ≤ 30s.

  * Subject, having given freely and expressly his/her informed consent.
  * Subject who is able to comply with the study requirements, as defined in the present CIP, at the Investigator's appreciation.
  * For applicable countries: subject being affiliated to a health social security system.
  * Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Far best corrected visual acuity < 1/10 (according to Snellen Chart)
* Subject with severe ocular dryness with one of these conditions:

  * Eyelid or blinking malfunction
  * Corneal disorders not related to dry eye syndrome
  * Ocular metaplasia
  * Filamentous keratitis
  * Corneal neovascularization
* Subject with severe meibomian gland dysfunction (MGD).
* History of ocular trauma, infection or inflammation, not related to dry eye syndrome within the last 3 months prior to the inclusion.
* History of ocular allergy or ocular herpes within the last 12 months.
* Any troubles of the ocular surface not related to dry eye syndrome .
* Subjects who underwent ocular surgery, including laser surgery, in either eye within the last 6 months.
* Use of the following ocular treatments: isotretinoïd, cyclosporine, tacrolimus, sirolimus, pimecrolimus, punctual plugs during the month preceding the inclusion.
* Subjects who have received ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start or expected to receive ocular therapy during the study.
* Any not stabilised systemic treatment, which can have an effect on performance or safety criteria, at the investigator appreciation.
* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject deprived of freedom by administrative or legal decision.
* Subject in a social or health institution.
* Subject who is under guardianship or who is not able to express his/her consent.
* Subject being in an exclusion period for a previous study.
* Subject suspected to be non-compliant according to the Investigator's judgment.
* Subject wearing contact lenses during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Cornea and conjunctiva staining (Oxford score) | 35 days
  Evaluation of the non-inferiority of DM934 in comparison with Théalose, in terms of cornea and conjunctiva staining (Oxford score), on worse eye

SECONDARY OUTCOMES:
Cornea and conjunctiva staining (Oxford score) (performance) | 35 days
  Main change from baseline of cornea and conjunctiva staining (Oxford score) in the worse eye and contralateral eye
Cornea and conjunctiva staining (Oxford score) (performance) | 84 days
  Main change from baseline of cornea and conjunctiva staining (Oxford score) in the worse eye and contralateral eye
Tear-Film Break Up Time (TBUT) (performance) | 35 days
  Main change from baseline of Tear-Film Break Up Time (TBUT) in the worse eye and contralateral eye
Tear-Film Break Up Time (TBUT) (performance) | 84 days
  Main change from baseline of Tear-Film Break Up Time (TBUT) in the worse eye and contralateral eye
OSDI (questionnaire)(performance) | 35 days
  Main change from baseline of Ocular Surface Disease Index (OSDI) score
OSDI (questionnaire)(performance) | 84 days
  Main change from baseline of Ocular Surface Disease Index (OSDI) score
Van Bijsterveld score (performance) | 35 days
  Main change from baseline of Van Bijsterveld score (lissamine green staining) in the worse eye and contralateral eye
Van Bijsterveld score (performance) | 84 days
  Main change from baseline of Van Bijsterveld score (lissamine green staining) in the worse eye and contralateral eye
Schirmer test (performance) | 35 days
  Main change from baseline of Schirmer test result in the worse eye and contralateral eye
Schirmer test (performance) | 84 days
  Main change from baseline of Schirmer test result in the worse eye and contralateral eye
Dry eye symptoms (performance) | 35 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D84 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Dry eye symptoms (performance) | 84 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D84 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Global performance by the investigator (performance) | 35 days
  Global performance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the investigator (performance) | 84 days
  Global performance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the patient (performance) | 35 days
  Global performance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the patient (performance) | 84 days
  lobal performance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Number of Adverse Events (safety) | 84 days
  Collection of ocular and systemic adverse events

OTHER OUTCOMES:
Lacrimal meniscus height (exploratory, optional) | 35 days
  Main change from baseline of lacrimal meniscus height in the worse eye and contralateral eye
Lacrimal meniscus height (exploratory, optional) | 84 days
  Main change from baseline of lacrimal meniscus height in the worse eye and contralateral eye

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Paw, MD, Principal Investigator — Eurofins Dermscan Poland
Locations (5):
- France (2):
  - Eurofins Dermscan, Aix-en-Provence
  - Eurofins EVIC, Bordeaux
- Eurofins Dermscan Poland, Gdansk, Poland
- IOBA, Valladolid, Spain
- Ocular Technology Group, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Depending on any journal publication of the results